CLINICAL TRIAL: NCT05763082
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Padagis' Roflumilast Cream 0.3% to Arcutis's Zoryve™ (Roflumilast Cream 0.3%) Cream and Both Active Treatments to a Vehicle Control in the Treatment of Plaque Psoriasis
Brief Title: Bioequivalence Study of Two Treatments for the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAD-NY-22-05
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Padagis active product (Experimental)
  Interventions: Drug: roflumilast cream 0.3%
- Reference product (Active Comparator)
  Interventions: Drug: Zoryve
- Padagis placebo product (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: roflumilast cream 0.3% — test product
  Arms: Padagis active product
Drug: Zoryve — Reference Listed Drug product
  Arms: Reference product
Drug: Placebo — placebo
  Arms: Padagis placebo product

SUMMARY:
To compare the safety and efficacy of Padagis' product to an FDA approved product for the treatment of plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Signed IRB approved written informed consent/assent
2. 12 to 75 years of age, inclusive.
3. Subjects must have a clinical diagnosis of stable symptomatic plaque psoriasis.
4. Baseline Investigator's Global Assessment Score of 3 (moderate).
5. Subjects must have a Body Surface Area (BSA) between 2% to 20%
6. Females of child bearing potential (excluding women who are surgically sterilized (tubal ligation or bilateral oophorectomy or hysterectomy) or post-menopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day1(Baseline), must be willing to use an acceptable form of birth control during the study.

Exclusion Criteria:

1. Pregnant, breastfeeding or planning a pregnancy within the period of their study participation period.
2. Current diagnosis of unstable forms of psoriasis in the treatment area.
3. History of unresponsiveness to topical treatment for psoriasis
4. Presence of any other skin condition that, in the Investigator's opinion, might interfere with psoriasis diagnosis and/or evaluations
5. Any uncontrolled, chronic or serious disease or medical condition that would prevent participation in a clinical trial, or, in judgment of the investigator, would put the subject at undue risk or might confound the study assessments
6. Use of medicated make-up throughout the study and significant change in the use of consumer products within 30 days (1 month) of study entry and throughout the study
7. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements.
8. Subjects who in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) | Day 1 to Day 56
  percentage of subjects at Day 56 who achieve Treatment Success, which is defined as an IGA score of None (0) or Minimal (1) with a 2-grade improvement from Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- DS Research, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No